CLINICAL TRIAL: NCT04053777
Title: Establishment and Validation of the Clinical Assessment Method in Patients Using Non-invasive Ventilation
Brief Title: Clinical Assessment Method in Patients Using Non-invasive Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guan Lili, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: GIRH-NIV201906
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NIV group: Patients receiving non-invasive ventilation in the hospital or at home
  Interventions: Device: non-invasive ventilation

INTERVENTIONS:
Device: non-invasive ventilation — Noninvasive positive pressure ventilation used assist/control mode to treat chronic respiratory disease.

SUMMARY:
This is an observational study of recording the respiratory parameters of patients when receiving non-invasive ventilation and analyze the relationship between those parameters and clinical outcomes.

DETAILED DESCRIPTION:
Non-invasive positive pressure ventilation (NPPV) is undoubtedly one of the most important advances in mechanical ventilation technology in the past 30 years. Currently, NPPV has become an essential respiratory support technology in hospitals, and it is used in different fields, including respiratory and critical care, emergency care, anesthesia, and rehabilitation. Applications of NPPV are also gradually expanding from intensive care units (ICUs) and respiratory wards to use in other medical departments and at home.

This is an observational study of recording the respiratory parameters of patients when receiving non-invasive ventilation and analyze the relationship between those parameters and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80, males and females
2. Patients with hypercapnic respiratory failure
3. Willing to participate in the study.
4. Being able to provide informed consent.

Exclusion Criteria:

1. Subjects with severe heart failure, severe arrhythmias, unstable angina, and malignant comorbidities.
2. Subjects with significantly impaired cognitive function and are unable to fulfill the study requirement (unable to provide informed consent)
3. Subjects who participated in another trial within 30 days prior to the planned start of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypercapnic respiratory failure who need to use non-invasive ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Changes of visual analogue scale score before and after using non-invasive ventilation | 1 hour
  Visual analogue scale score is used to represent the subjective dyspnea of patient. Scores range between 0 and 10 and higher scores are attributed to less dyspnea.

SECONDARY OUTCOMES:
Changes of respiratory rate before and after using non-invasive ventilation | 1 hour
  The respiratory rate is the rate at which breathing occurs. This is usually measured in breaths per minute.
Changes of SpO2 before and after using non-invasive ventilation | 1 hour
  Oxygen saturation is the fraction of [oxygen]-saturated hemoglobin relative to total hemoglobin in the blood.
Changes of tidal volume before and after using non-invasive ventilation | 1 hour
  Tidal volume is the lung volume representing the normal volume of air displaced between normal inhalation and exhalation when extra effort is not applied.This is usually measured in mini Liter.
Changes of heart rate before and after using non-invasive ventilation | 1 hour
  Heart rate is the speed of the heartbeat measured by the number of contractions (beats) of the heart per minute (bpm).

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China